CLINICAL TRIAL: NCT01870921
Title: A Multicenter, Single Arm, Open Label, Phase IV Study to Evaluate Safety and to Describe the Incidence of Major Cardiovascular Events of Ticagrelor in Chinese Patients With Acute Coronary Syndrome(ACS)
Brief Title: Brilinta DaYu Study
Acronym: DaYu
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D5130C00087
Record Dates: First submitted 2013-06-04; First posted 2013-06-06 (Estimated); Results first posted 2016-11-09 (Estimated); Last update posted 2018-04-03 (Actual); Status verified 2018-03

CONDITIONS: Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Ticagrelor

ARMS (1):
- Ticargrelor (Experimental): 90 mg/tablet, 1 tablet bid
  Interventions: Drug: Ticagrelor

INTERVENTIONS:
Drug: Ticagrelor — 90mg/tablet, 1 tablet bid

SUMMARY:
A multicenter, single arm, open label, Phase IV study to evaluate safety and to describe the incidence of major cardiovascular events of ticagrelor in Chinese patients with acute coronary syndrome

ELIGIBILITY:
Inclusion Criteria:

* 1. Female or male aged at least 18 years 2.Index event of non-ST or ST segment elevation ACS 3.A patient who is considered as ethnic Chinese

Exclusion Criteria:

* 1. With coagulation disorder 2.Index event is an acute complication of PCI 3.Patient has planned for an urgent coronary artery bypass graft (CABG) within 7days from the enrolment 4.Oral anticoagulation therapy within 30 days prior to enrolment or cannot be stopped 5.Increased risk of bradycardic events 6. Concomitant oral or intravenous therapy (see examples below) with strong CYP3A inhibitors, CYP3A substrates with narrow therapeutic indices, or strong CYP3A inducers 7.Increased risk of bradycardic events (eg, no pacemaker and known sick sinus syndrome, second degree A-V block, third degree A-V block or previous documented syncope suspected to be due to bradycardia unless treated with a pacemaker). 8.Known clinically important thrombocytopenia 9.Known clinically important anaemia

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2004 (Actual)
Dates: Start 2013-06-26 (Actual); Primary Completion 2015-09-30 (Actual); Study Completion 2015-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Runlin Gao, Doctor, Principal Investigator — Fu Wai Hospital, Beijing, China
Locations (21):
- China (21):
  - Research Site, Beijing
  - Research Site, Changchun
  - Research Site, Chengdu
  - Research Site, Chuangchun
  - Research Site, Fuzhou
  - Research Site, Guangzhou
  - Research Site, Jinan
  - Research Site, Jining
  - Research Site, Kunming
  - Research Site, Nanjing
  - Research Site, Shanghai
  - Research Site, Shenyang
  - Research Site, Shenzhen
  - Research Site, Taiyuan
  - Research Site, Wuhan
  - Research Site, Wuxi
  - Research Site, Xi'an
  - Research Site, Xiamen
  - Research Site, Xuzhou
  - Research Site, Zhengzhou
  - Research Site, Zhongshan

REFERENCES:
- [Background] Gao R, Wu Y, Liu H, Su G, Yuan Z, Zhang A, Wang Y, Wang Z, Wang Y, Zhang H, Zheng Y, Liu L, Shen L, Leonsson-Zachrisson M, Han Y; DAYU study investigators. Safety and Incidence of Cardiovascular Events in Chinese Patients with Acute Coronary Syndrome Treated with Ticagrelor: the 12-Month, Phase IV, Multicenter, Single-Arm DAYU Study. Cardiovasc Drugs Ther. 2018 Feb;32(1):47-56. doi: 10.1007/s10557-018-6772-3. PMID 29488142
- See also: D5130C00087 Clinical Study Protocol and amendment redacted — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1829&filename=D5130C00087%20_Clinical%20StudyProtocol_and_amendment_redacted.pdf

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ticargrelor
Started | 2004
Completed | 1914
Not Completed | 90
Not completed — Subject decision | 80
Not completed — Severe non-compliance to protocol | 7
Not completed — Subject Lost to Follow up | 2
Not completed — Other | 1

BASELINE CHARACTERISTICS:
Population: Based on the safety population, i.e. all enrolled patients who received at least one dose of Investigational product (IP)
Arm/Group | Ticargrelor
Number analyzed (Participants) | 2001
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.3 (10.83)
Age, Customized [Number; unit: Participants]
  < 75 years | 1854
  >= 75 years | 147
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 422
  Male | 1579
Race/Ethnicity, Customized [Number; unit: Participants] — Ethnic Group
  Participants
    Hispanic or latino | 0
    Not hispanic or latino | 2001
Race/Ethnicity, Customized [Number; unit: Participants] — Race
  Participants
    Asian | 2001
    Other | 0

OUTCOME MEASURES:

1. Primary Outcome: Bleeding Events
Description: PLATO-defined fatal/life threatening, major, major+minor,major+minor+minimal
Time Frame: 12 months
Measure: Number; unit: Participants
Arm/Group | Ticargrelor
Number analyzed (Participants) | 2001
Participants
  Fatal/life threatening | 17
  Major | 27
  Major + minor | 93
  Major + minor + minimal | 426

2. Primary Outcome: Serious Adverse Events Other Than Bleeding
Description: SAEs except the blending events which have aleady been reported as SAEs.
Time Frame: 12 months
Measure: Number; unit: Participants
Arm/Group | Ticargrelor
Number analyzed (Participants) | 2001
Participants | 116

3. Secondary Outcome: Major CV Events
Description: Combination of CV death, MI, and stroke
Time Frame: 12 months
Measure: Number; unit: Participants
Arm/Group | Ticargrelor
Number analyzed (Participants) | 2001
Participants | 85

ADVERSE EVENTS:
Time Frame: From day of first dose to the day of last dose + 7 days, up to 1 year.
Arm/Group | Ticargrelor
Serious Adverse Events (participants affected / at risk) | 161/2001
Other Adverse Events (participants affected / at risk) | 230/2001
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ticargrelor (N=2001)
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 16 (16)
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 12 (12)
Gastritis (Gastrointestinal disorders) | 4 (5)
Duodenal Ulcer Haemorrhage (Gastrointestinal disorders) | 3 (3)
Gastric Ulcer Haemorrhage (Gastrointestinal disorders) | 2 (2)
Faeces Discoloured (Gastrointestinal disorders) | 1 (1)
Gastritis Erosive (Gastrointestinal disorders) | 1 (1)
Gingival Bleeding (Gastrointestinal disorders) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 1 (1)
Inguinal Hernia (Gastrointestinal disorders) | 1 (1)
Intestinal Obstruction (Gastrointestinal disorders) | 1 (1)
Cardiac Failure (Cardiac disorders) | 5 (5)
Acute Left Ventricular Failure (Cardiac disorders) | 3 (3)
Cardiac Failure Chronic (Cardiac disorders) | 3 (3)
Angina Pectoris (Cardiac disorders) | 1 (1)
Angina Unstable (Cardiac disorders) | 1 (1)
Arrhythmia (Cardiac disorders) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 1 (1)
Cardiac Failure Acute (Cardiac disorders) | 1 (1)
Cardiac Failure Congestive (Cardiac disorders) | 1 (1)
Cardio-Respiratory Arrest (Cardiac disorders) | 1 (1)
Coronary Artery Disease (Cardiac disorders) | 1 (1)
Coronary Artery Thrombosis (Cardiac disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Pericardial Effusion (Cardiac disorders) | 1 (1)
Sinus Arrest (Cardiac disorders) | 1 (1)
Ventricular Arrhythmia (Cardiac disorders) | 1 (1)
Ventricular Septal Defect Acquired (Cardiac disorders) | 1 (1)
Lung Infection (Infections and infestations) | 4 (4)
Pneumonia (Infections and infestations) | 3 (3)
Appendicitis (Infections and infestations) | 2 (2)
Urinary Tract Infection (Infections and infestations) | 2 (2)
Cystitis (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
Lower Respiratory Tract Infection (Infections and infestations) | 1 (1)
Pneumonia Klebsiella (Infections and infestations) | 1 (1)
Pulmonary Tuberculosis (Infections and infestations) | 1 (1)
Respiratory Tract Infection (Infections and infestations) | 1 (1)
Septic Shock (Infections and infestations) | 1 (1)
Upper Respiratory Tract Infection (Infections and infestations) | 1 (1)
Chronic Kidney Disease (Renal and urinary disorders) | 4 (4)
Haematuria (Renal and urinary disorders) | 4 (4)
Haemorrhage Urinary Tract (Renal and urinary disorders) | 1 (1)
Hypertensive Nephropathy (Renal and urinary disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1)
Renal Artery Stenosis (Renal and urinary disorders) | 1 (1)
Renal Failure (Renal and urinary disorders) | 1 (1)
Cerebral Haemorrhage (Nervous system disorders) | 4 (4)
Subarachnoid Haemorrhage (Nervous system disorders) | 3 (3)
Cerebral Infarction (Nervous system disorders) | 1 (1)
Hypoglycaemic Coma (Nervous system disorders) | 1 (1)
Intercostal Neuralgia (Nervous system disorders) | 1 (1)
Neuropathy Peripheral (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Chest Discomfort (General disorders) | 6 (6)
Sudden Death (General disorders) | 3 (3)
Multi-Organ Failure (General disorders) | 1 (1)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Bronchitis Chronic (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 4 (4)
Gouty Arthritis (Musculoskeletal and connective tissue disorders) | 2 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Road Traffic Accident (Injury, poisoning and procedural complications) | 2 (2)
Brain Contusion (Injury, poisoning and procedural complications) | 1 (1)
Injury (Injury, poisoning and procedural complications) | 1 (1)
Skin Abrasion (Injury, poisoning and procedural complications) | 1 (1)
Soft Tissue Injury (Injury, poisoning and procedural complications) | 1 (1)
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 1 (1)
Vascular Pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1)
Diabetes Mellitus Inadequate Control (Metabolism and nutrition disorders) | 4 (5)
Type 2 Diabetes Mellitus (Metabolism and nutrition disorders) | 2 (2)
Gout (Metabolism and nutrition disorders) | 1 (1)
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Bronchial Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Gastric Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastatic Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Myeloproliferative Disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Arteriovenous Fistula (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Peripheral Arterial Occlusive Disease (Vascular disorders) | 1 (1)
Peripheral Venous Disease (Vascular disorders) | 1 (1)
Subclavian Artery Stenosis (Vascular disorders) | 1 (1)
Orthostatic Hypotension (Vascular disorders) | 1 (1)
Cholecystitis Acute (Hepatobiliary disorders) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1)
Hepatic Function Abnormal (Hepatobiliary disorders) | 1 (1)
Liver Disorder (Hepatobiliary disorders) | 1 (1)
Depression (Psychiatric disorders) | 2 (2)
Completed Suicide (Psychiatric disorders) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Haemolytic Anaemia (Blood and lymphatic system disorders) | 1 (1)
Aural Polyp (Ear and labyrinth disorders) | 1 (1)
Middle Ear Inflammation (Ear and labyrinth disorders) | 1 (1)
Vertigo Positional (Ear and labyrinth disorders) | 1 (1)
Primary Hyperaldosteronism (Endocrine disorders) | 1 (1)
Thyroid Mass (Endocrine disorders) | 1 (1)
Blindness Unilateral (Eye disorders) | 1 (1)
Cataract (Eye disorders) | 1 (1)
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 1 (1)
Cervical Polyp (Reproductive system and breast disorders) | 1 (1)
Drug Hypersensitivity (Immune system disorders) | 1 (1)
Blood Glucose Increased (Investigations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ticargrelor (N=2001)
Ecchymosis (Skin and subcutaneous tissue disorders) | 113 (130)
Hyperuricaemia (Metabolism and nutrition disorders) | 130 (132)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At least sixty (60) days prior to submission of any material for publication or presentation, Institution shall provide AstraZeneca with such material for review. If requested in writing by AstraZeneca, Institution shall withhold material from submission for publication or presentation for an additional ninety (90) days to allow for the filing of a patent application or the taking of such measures as AstraZeneca deems appropriate to establish and preserve its proprietary rights.